CLINICAL TRIAL: NCT04423250
Title: Pilot Study Evaluating the Impact of the Intervention of a Pharmacist in the Operating Room on the Appropriate Use of Sterile Medical Devices and the Economic Repercussions
Brief Title: Evaluating the Impact of the Intervention of a Pharmacist in the Operating Room on the Appropriate Use of Sterile Medical DeviceS
Acronym: OPTIBLOC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2016/JMK-01
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: impact of the intervention of a clinical pharmacist with expertise in sterile medical devices on non-compliances related to the use of sterile medical devices — - Failure to trace, Lack of product information, absence of product in the operating room

SUMMARY:
assess the impact of the intervention of a clinical pharmacist expert in sterile medical devices

ELIGIBILITY:
Inclusion Criteria:

* - The patient must be a member or beneficiary of a health insurance plan.
* The patient is managed for scheduled surgery (full hospitalization or outpatient) in the UDG (Urology Digestive Gynecology) operating room.

Exclusion Criteria:

* - The subject is in a period of exclusion determined by a previous study.
* The subject is under judicial protection.
* The subject (or his/her legal representative) has expressed his/her opposition to participate in the study.
* The patient is undergoing emergency surgery in the UDG (Urology Digestive Gynecology) operating room.
* It is not possible to give informed information about the subject.

Translated with www.DeepL.com/Translator (free version)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for scheduled surgery in the UDG (Urology Digestive Gynecology) operating room.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
identify compliance with the appropriate use of sterile medical devices | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No